CLINICAL TRIAL: NCT03919149
Title: Psychological and Social Determinants of Physical Activity Practice From Diagnose to Survival Among French Cancer Patients
Brief Title: Psycho-social Determinant for Sport Practised During Cancer
Acronym: PERTINENCE
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-08Obs-CHRMT
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Cancer
MeSH Terms: conditions — Motor Activity; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The litterature has demonstrates that physical activity can play an important role in decreasing patient mortality rates and increasing its well-being at all time of cancer. Despite this evidence, there is a weak adhesion in patients. It is therefore appropriate to look and see which may explain the high prevalence of physical inactivity in patients with cancer. The main objective of this study will be to recognize psychological and social factors which could explain the commitment or not to a physical activity in cancer patients. Besides the physical limitations related to the cancer and its treatment, socio-economic and psycho-social factors can often play an extremely important role in engagement or maintenance of sporting activity.

DETAILED DESCRIPTION:
Different individual factors have been identified as playing an important role in physical activity (PA) practice. For example, sex, age, education level, socio-professional category, ethnicity, overweight seemed to impact PA level in general population and among cancer patient.

Beyond the disease's effect, as well as its treatment, the socio-ecological approach has identified five group of factors associated to PA practice: individual factors, interpersonal factors, environmental factors, political factors and global factors.

The aim of this mixed methods study is to identify the variables of the socioecological model facilitating PA practice, as well as PA level and preferences at different time during cancer (at diagnose, during treatment, after treatment).

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* With an histollogically confirmed non-metastatic (breast, prostate or colorectal) cancer diagnosis
* To be addressed to an oncologist before the beginning of any treatment
* Informed and having agreed to participate in the study
* Operated patient without adjuvant therapy

Exclusion Criteria:

* Presence of threatening bone lesion
* physical, cognitive or linguistics incapacity to fulfil the questionnaire
* With a life expectancy of less than 6 months
* Pregnant woman
* Under legal protection or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an histollogically confirmed non-metastatic breast, prostate or colorectal cancer diagnosis, who had no started any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Physical activity | Day 1
  The Questionnaire include four main section: medical, socio-economic variables, personality traits situational variables and physical activity. Sociological variables will encompass age, gender, education, and socio-professional category, and professional activity, marital and socio-economic status, place of living. Life habits and PA practice before diagnose will help to look at inter-determinants relationships. Medical data will also be collected from patient perspective. Situational variables will encompass passion, basic need satisfaction in sport, state-hope, self-determined motivation for PA, anxiety and depression. PA and sedentary behaviors will be measured using self-reported Global Physical Activity questionnaire. This questionnaire will measure the frequency, intensity, duration, as well as context of PA practice.

SECONDARY OUTCOMES:
Physical activity at 6 months | Month 6
  The Questionnaire six months after the inclusion
Physical activity at 12 months | Month 12
  The Questionnaire one year after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Tarquino Cyril, Pr, Study Chair — Centre Pierre Janet, Université de Lorraine
Locations (3):
- France (3):
  - CHR Metz Thionville, Metz
  - Institut de Cancérologie de Lorraine, Nancy
  - CHR Metz Thionville, Thionville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Hoye A, Omorou Y, Rotonda C, Gendarme S, Tarquinio C, Houtmann B, Peiffert D, Longo R, Martin-Krumm C. Psychological and social determinants of physical activity from diagnosis to remission among French cancer patients (PERTINENCE): protocol for a mixed-method study. BMC Public Health. 2019 Aug 6;19(1):1053. doi: 10.1186/s12889-019-7368-y. PMID 31387577